CLINICAL TRIAL: NCT00001318
Title: Treatment of Non-Tuberculous Mycobacterial Infections With Interferon Gamma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920255; 92-I-0255
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Healthy; Mycobacterium Infections, Atypical
Keywords: Immune Adjuvant; Phagocytes; Non-tuberculous Mycobacterial Infection
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Interferon-gamma

INTERVENTIONS:
Drug: interferon gamma

SUMMARY:
This is an open label study to determine the effects of the administration of Interferon-gamma on the clinical condition and immune function of patients with severe, treatment refractory non-tuberculosis mycobacterial infections. The study drug (interferon gamma) will be administered subcutaneously three times a week at 0.05 mg/m(2) for one year. We may also collect blood from the relatives of these patients and normal volunteers in order to characterize the genetic basis, if any, of our patients' disorders.

DETAILED DESCRIPTION:
This is an open label study to determine the effects of the administration of Interferon-gamma on the clinical condition and immune function of patients with severe, treatment refractory non-tuberculosis mycobacterial infections. The study drug (interferon gamma) will be administered subcutaneously three times a week at 0.05 mg/m(2) for one year. We may also collect blood from the relatives of these patients and normal volunteers in order to characterize the genetic basis, if any, of our patients' disorders.

ELIGIBILITY:
Demonstrated non-tuberculous mycobacterial infection, either disseminated or pulmonary.

Received medical treatment for at least 3 months without improvement.

Preserved renal, hepatic and hematologic function.

Negative pregnancy urine and effective contraceptive.

Age range greater than 5.

No secondary immunodeficiency such as HIV or malignancy.

Not currently receiving cytotoxic therapy within the past 3 months.

Not pregnant or lactating.

No seizure disorders.

No known symptomatic cardiac disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1992-08; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nathan CF, Kaplan G, Levis WR, Nusrat A, Witmer MD, Sherwin SA, Job CK, Horowitz CR, Steinman RM, Cohn ZA. Local and systemic effects of intradermal recombinant interferon-gamma in patients with lepromatous leprosy. N Engl J Med. 1986 Jul 3;315(1):6-15. doi: 10.1056/NEJM198607033150102. PMID 3086725
- [Background] Horsburgh CR Jr, Mason UG 3rd, Farhi DC, Iseman MD. Disseminated infection with Mycobacterium avium-intracellulare. A report of 13 cases and a review of the literature. Medicine (Baltimore). 1985 Jan;64(1):36-48. doi: 10.1097/00005792-198501000-00003. PMID 3880852
- [Background] Holland SM, Eisenstein EM, Kuhns DB, Turner ML, Fleisher TA, Strober W, Gallin JI. Treatment of refractory disseminated nontuberculous mycobacterial infection with interferon gamma. A preliminary report. N Engl J Med. 1994 May 12;330(19):1348-55. doi: 10.1056/NEJM199405123301904. PMID 7908719